CLINICAL TRIAL: NCT05295810
Title: Investigating Hypercapnia to Treat Neurogenic Orthostatic Hypotension
Brief Title: Hypercapnia in Orthostatic Hypotension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Satish Raj, Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB20-1322
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Orthostatic Hypotension; Neurogenic Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: Male and female NOH patients (n=40) will be recruited from the Calgary Autonomic Clinic, along with sex and age-matched controls from the community. Participants will complete five Active Stand Tests during which they will be asked to target different end-tidal (ET) CO2 levels. Participants will complete the following breathing protocol during an active stand test:
  1. Breathing normal room air (ETCO2 free to fluctuate),
  2. ETCO2 clamped at baseline,
  3. ETCO2 clamped at +5mmHg,
  4. ETCO2 clamped at +10mmHg,
  5. ETCO2 clamped at +10mmHg with ETO2 clamped at 50mmHg.
Masking Description: All participants will be fitted with a face mask connected to a tube supplied with gas from the RespirAct™ system. The participants will not be informed about the concentration of gases during each active stand test. After the study completion they will be informed about the order of interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Room Air (No Intervention): All participants will complete an active stand breathing room air with CO2 free to fluctuate
- +0mmHg CO2 Clamped at baseline (Experimental): All participants will complete an active stand with their CO2 held constant at baseline
  Interventions: Drug: Sequential Gas Delivery
- +5mmHg CO2 (Experimental): All participants will complete an active stand breathing +5mmHg of CO2 relative to baseline
  Interventions: Drug: Sequential Gas Delivery
- +10mmHg (Experimental): All participants will complete an active stand breathing +10mmHg of CO2 relative to baseline
  Interventions: Drug: Sequential Gas Delivery
- +10mmHg CO2 + 50mmHg O2 (Experimental): All participants will complete an active stand breathing +10mmHg of CO2 relative to baseline and 50mmHg of O2
  Interventions: Drug: Sequential Gas Delivery

INTERVENTIONS:
Drug: Sequential Gas Delivery — Sequential Gas Delivery will be controlled using the RespirAct™ system (Thornhill Research Inc., Toronto, Canada)
  Arms: +0mmHg CO2 Clamped at baseline; +10mmHg; +10mmHg CO2 + 50mmHg O2; +5mmHg CO2

SUMMARY:
The Autonomic (or "automatic") Nervous System (ANS) regulates internal processes, including control of heart rate and blood pressure (BP). When someone stands, and gravity tries to pull blood away from the brain, the ANS works to maintain BP and brain blood flow. Neurogenic Orthostatic Hypotension (NOH) occurs when our "fight-or-flight" part ("sympathetic") of the ANS fails. BP can drop a lot when upright, reducing blood flow and oxygen delivery to the brain, and this can cause symptoms of light-headedness, nausea, and fainting.

One solution to help counter the effects of NOH may be to increase sympathetic activity by breathing higher levels of carbon dioxide. In healthy volunteers, small increases in the amount of inhaled carbon dioxide has been shown to increase BP in the upright position, and this improves symptoms!

The objectives of the current study are to apply carbon dioxide in patients with NOH and healthy controls to: (a) evaluate the effects of breathing carbon dioxide on BP and brain blood flow, and (b) determine if a device that increases carbon dioxide while standing will work as a new therapy

DETAILED DESCRIPTION:
BACKGROUND: Regulation of tissue blood supply to vital organs such as the brain and heart is met in large part by local adjustment of the microvasculature (autoregulation) and autonomic nervous system control of the cardiovascular system. Neurogenic Orthostatic Hypotension (NOH) is a key example of when these systems fail. Patients experience a significant and persistent blood pressure (BP) drop (≥20/10 mmHg) in the upright position, resulting in cerebral hypoperfusion and symptoms of light-headedness, nausea, pre-syncope and even syncope. NOH and impaired cerebrovascular perfusion occur due to failure of the baroreflex to appropriately increase sympathetic outflow.

A novel solution to counter the acute effects of NOH is to transiently increase sympathetic activity by stimulating the peripheral and central respiratory chemoreceptors with elevated Fractional Inspired (Fi)CO2. In healthy volunteers, elevated FiCO2 improves orthostatic tolerance and BP control during rapid postural transitions. Additionally, few have considered sex-difference effects on the chemoreflex-autonomic relationship. Existing evidence demonstrates an augmented sympathetic response to chemoreflex stimulation in postmenopausal women with observed vasoconstriction and increased BPs. These data indicate females may respond better to hypercapnia as a novel therapeutic intervention for NOH. Unfortunately, it may also highlight a predisposition for cardiovascular risk associated with supine hypertension.

To better understand the mechanistic underpinnings of NOH in males and females, and to explore the use of elevated FiCO2 to treat it, researchers need a better way to monitor sympathetic activity and cerebrovascular perfusion. Functional Optical Coherence Tomography (fOCT) of the retinal and choroid vascular beds of the eye (an out crop of the brain) was recently developed in Calgary to allow physiological monitoring of these essential variables. In summary, elevated FiCO2 levels (hypercapnia) appear to improve BP responses to standing and orthostatic tolerance and may constitute an attractive therapy for NOH patients.

This is a proof-of-concept study to evaluate hypercapnia as a novel therapeutic intervention to improve blood pressure and orthostatic tolerance in male and female patients with NOH. In addition, the investigators will aim to evaluate functional OCT as an advance, non-invasive tool to measure sympathetic and metabolic cerebrovascular control.

OBJECTIVES: The aims of the current proposal are to apply hypercapnia during fOCT monitoring in male and female patients with NOH and healthy controls to: (a) evaluate and compare the effects of hypercapnia on cardiovascular and cerebrovascular responses to better understand basic chemoreflex and baroreflex physiology in male and female patients with NOH, (b) determine if a device that transiently increases FiCO2 in response to postural changes will have efficacy as a non-drug therapeutic and (c) evaluate fOCT as a novel advanced tool to measure sympathetic and metabolic components of cerebral autoregulation in patients with autonomic failure.

METHODS: Male and female NOH patients (n=40) will be recruited from the Calgary Autonomic Clinic, along with sex and age-matched controls from the community. Participants will complete five Active Stand Tests during which they will be asked to target different end-tidal (ET) CO2 levels. OCT images will be captured throughout each test. Participants will complete the following breathing protocol during an active stand test: a) breathing normal room air (ETCO2 free to fluctuate), b) ETCO2 clamped at baseline, c) ETCO2 clamped at +5mmHg, d) ETCO2 clamped at +10mmHg, e) ETCO2 clamped at +10mmHg with ETO2 clamped at 50mmHg. Target ETCO2 levels will be achieved through a computerized gas delivery system. A rebreathing task to elicit hypercapnia and hypoxia (low oxygen) will be performed last. Each condition will be followed by a minimum 10-minute recovery period to ensure ETCO2 normalization. Hemodynamics (BP, HR and stroke volume) and orthostatic symptoms will be assessed throughout. Breath-by-breath data will include ETO2, ETCO2, respiration rate, tidal volume, and minute ventilation. OCT image analyses in the seated and standing position will measure choroid and retinal (surrogates for peripheral sympathetic activity and metabolic cerebral autoregulation, respectively) perfusion densities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Male and Female
* Non - smokers.
* Able and willing to provide informed consent.
* Ability to travel to Libin Cardiovascular Institute Autonomic Testing Lab at the University of Calgary, Calgary, AB.

Exclusion Criteria:

* Medical therapies or medications which could interfere with testing of autonomic function
* Participants with somatization or severe anxiety symptoms will be excluded
* Pregnant or breast-feeding females
* Inability to tolerate mask for the duration of the study
* Subjects who require portable oxygen at rest or with exercise
* Subjects with chronic heart failure or severe pulmonary disease who are unable to climb one flight of stairs due to shortness of breath.
* Presence of failure of other organ systems or systemic illness that can affect autonomic function or the participant's ability to cooperate. These include: dementia, alcohol and/or drug abuse, cerebrovascular disease, kidney or liver disease, surgical procedures where the nerves of the sympathetic nervous system have been cut.
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Δ Blood Pressure (BP) | The ΔBP (stand-sit) calculated as the average BP in the final minute of sitting and the average BP between minute 3 and 5 of stand will be compared between room air and +10mmHg of CO2
  Magnitude of ΔBP (Stand-Sit) breathing room air vs +10mmHg of CO2

SECONDARY OUTCOMES:
Δ Blood Pressure (BP) | The ΔBP (stand-sit) calculated as the average BP in the final minute of sitting and the average BP between minute 3 and 5 of stand will be compared between room air and 0 mmHg of CO2
  Magnitude of ΔBP (Stand-Sit) breathing room air vs 0 mmHg of CO2
Δ Blood Pressure (BP) | The ΔBP (stand-sit) calculated as the average BP in the final minute of sitting and the average BP between minute 3 and 5 of stand will be compared between room air and +5mmHg of CO2
  Magnitude of ΔBP (Stand-Sit) breathing room air vs +5mmHg of CO2
Δ Blood Pressure (BP) | The ΔBP (stand-sit) calculated as the average BP in the final minute of sitting and the average BP between minute 3 and 5 of stand will be compared between room air and +10mmHgCO2/50mmHg O2
  Magnitude of ΔBP (Stand-Sit) breathing room air vs +10mmHgCO2/50mmHg O2
Δ Vanderbilt Orthostatic Symptom Score [Range: 0 (absent) to 10 (worst)] | The Δ Vanderbilt Orthostatic Symptom Score (symptoms at the 5th minute of stand - symptoms at the 5th minute of sit) will be compared between room air and +10mmHg of CO2
  Magnitude of Δ Vanderbilt Orthostatic Symptom Score (Stand-Sit) breathing room air vs +10mmHg of CO2
Δ Vanderbilt Orthostatic Symptom Score [Range: 0 (absent) to 10 (worst)] | The Δ Vanderbilt Orthostatic Symptom Score (symptoms at the 5th minute of stand - symptoms at the 5th minute of sit) will be compared between room air and 0 mmHg of CO2
  Magnitude of Δ Vanderbilt Orthostatic Symptom Score (Stand-Sit) breathing room air vs 0 mmHg of CO2
Δ Vanderbilt Orthostatic Symptom Score [Range: 0 (absent) to 10 (worst)] | The Δ Vanderbilt Orthostatic Symptom Score (symptoms at the 5th minute of stand - symptoms at the 5th minute of sit) will be compared between room air and +5mmHg of CO2
  Magnitude of Δ Vanderbilt Orthostatic Symptom Score (Stand-Sit) breathing room air vs +5mmHg of CO2
Δ Vanderbilt Orthostatic Symptom Score [Range: 0 (absent) to 10 (worst)] | The Δ Vanderbilt Orthostatic Symptom Score (symptoms at the 5th minute of stand - symptoms at the 5th minute of sit) will be compared between room air and +10mmHgCO2/50mmHg O2
  Magnitude of Δ Vanderbilt Orthostatic Symptom Score (Stand-Sit) breathing room air vs +10mmHgCO2/50mmHg O2
Δ Cerebral Blood Flow Velocity (CBFv) | The ΔCBFv (stand-sit) calculated as the average CBFv in the final minute of sitting and the average CBFv between minute 3 and 5 of stand will be compared between room air and +10mmHg of CO2
  Magnitude of ΔCBFv (Stand-Sit) breathing room air vs +10mmHg of CO2
Δ Cerebral Blood Flow Velocity (CBFv) | The ΔCBFv (stand-sit) calculated as the average CBFv in the final minute of sitting and the average CBFv between minute 3 and 5 of stand will be compared between room air and 0 mmHg of CO2
  Magnitude of ΔCBFv (Stand-Sit) breathing room air vs 0 mmHg of CO2
Δ Cerebral Blood Flow Velocity (CBFv) | The ΔCBFv (stand-sit) calculated as the average CBFv in the final minute of sitting and the average CBFv between minute 3 and 5 of stand will be compared between room air and +5mmHg of CO2
  Magnitude of ΔCBFv (Stand-Sit) breathing room air vs +5mmHg of CO2
Δ Cerebral Blood Flow Velocity (CBFv) | The ΔCBFv (stand-sit) calculated as the average CBFv in the final minute of sitting and the average CBFv between minute 3 and 5 of stand will be compared between room air and +10mmHgCO2/50mmHg O2
  Magnitude of ΔCBFv (Stand-Sit) breathing room air vs +10mmHgCO2/50mmHg O2

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Freeman R, Abuzinadah AR, Gibbons C, Jones P, Miglis MG, Sinn DI. Orthostatic Hypotension: JACC State-of-the-Art Review. J Am Coll Cardiol. 2018 Sep 11;72(11):1294-1309. doi: 10.1016/j.jacc.2018.05.079. PMID 30190008
- [Background] Morgan BJ, Crabtree DC, Palta M, Skatrud JB. Combined hypoxia and hypercapnia evokes long-lasting sympathetic activation in humans. J Appl Physiol (1985). 1995 Jul;79(1):205-13. doi: 10.1152/jappl.1995.79.1.205. PMID 7559221
- [Background] Schultz HD, Li YL, Ding Y. Arterial chemoreceptors and sympathetic nerve activity: implications for hypertension and heart failure. Hypertension. 2007 Jul;50(1):6-13. doi: 10.1161/HYPERTENSIONAHA.106.076083. Epub 2007 May 14. No abstract available. PMID 17502495
- [Background] Shoemaker JK, O'Leary DD, Hughson RL. PET(CO(2)) inversely affects MSNA response to orthostatic stress. Am J Physiol Heart Circ Physiol. 2001 Sep;281(3):H1040-6. doi: 10.1152/ajpheart.2001.281.3.H1040. PMID 11514269
- [Background] Howden R, Lightfoot JT, Brown SJ, Swaine IL. The effects of breathing 5% CO2 on human cardiovascular responses and tolerance to orthostatic stress. Exp Physiol. 2004 Jul;89(4):465-71. doi: 10.1113/expphysiol.2004.027250. Epub 2004 May 6. PMID 15131068

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT05295810/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT05295810/ICF_001.pdf